CLINICAL TRIAL: NCT03223064
Title: Accuracy of Lymph Node Imaging in Prostate Cancer: A Prospective Cohort Study to Determine the Concordance Between Two Imaging Modalities, "Combidex" Magnetic Resonance Imaging (Nano MRI) and 68Ga-PSMA Positron Emission Tomography (PET)
Brief Title: Accuracy of Lymph Node Imaging in Prostate Cancer: PSMA PET-CT and Nano-MRI
Acronym: MAGNIFY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry); Canisius-Wilhelmina Hospital (Other); Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ASTELLAS/MAGNIFY
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer; Lymph Node Metastases
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA PET-CT and USPIO MRI (Experimental)
  Interventions: Diagnostic Test: Ferumoxtran-10 enhanced MRI; MRI contrast agent; Diagnostic Test: 68Ga PSMA PET-CT

INTERVENTIONS:
Diagnostic Test: Ferumoxtran-10 enhanced MRI; MRI contrast agent — Patient undergo MRI with an USPIO contrast agent
Diagnostic Test: 68Ga PSMA PET-CT — Patient undergo an 68Ga PSMA PET-CT scan

SUMMARY:
Following curative intended therapy in prostate cancer patients, a high proportion of patients (approx. 25%) relapse with local and/or distant recurrence. The metastasis of a lymph node (LN) in a patient with prostate cancer means that the disease has become systemic with the increased risk of disease progression. Therefore the ability to detect the presence of LN metastasis is important in terms of disease prognosis and treatment options. In the past, patients with LN metastasis have had poor prognoses due to the scarcity of accurate staging techniques and toxic treatment regimens such as radiotherapy. For those patients with a medium to high risk of having LN metastasis, the current procedure is a bilateral pelvic lymph node dissection (PLND). This is the standard procedure prior to curative treatment with either radical prostatectomy or radiation therapy. However, the procedure is not optimal due to the frequent inability to remove all positive lymph nodes within the dissection area. 41% of metastatic LN disease is not found, due to these LN being outside the routine surgery field. As a result, some urologists will perform an extended lymphadenectomy (e-PLND), which leads to extended operating times and the risk of complications. Also, therapy of LN metastases has limitations: more than 50% of metastatic LN are outside the routine (RTOG-CTV) radiation field. Thus the effect of standard LN radiotherapy is limited. Currently used imaging techniques such as CT and conventional MRI are also not sensitive enough to detect prostate cancer metastases due to the small size of the nodes (< 8mm).

In this study, patients that undergo a pelvic lymph node dissection will be undergoing a 68Ga PSMA PET-CT and a nano-MRI prior to surgery. The results of the PSMA PET-CT and the nano-MRI will be validated using the pathology results of the (PLND).

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 years Prostate cancer present (Gleason ≥ 7) and/or
* PSA ≥ 15 and/or
* Clinical or radiological Stage T3
* Subject will be undergoing a pelvic lymph node dissection as part of the prostate cancer treatment.
* Subject is willing to sign and date the study Informed Consent form
* Signed, written informed consent

Exclusion Criteria:

* Patients who cannot lie still for at least 30 minutes or comply with imaging
* Subject has medical conditions that would limit study participation (per physician discretion)
* Subject has hemochromatosis and liver disease
* Subject has known allergy against Fe-products or dextranes
* Subject is enrolled in one or more concurrent studies that would confound the study results of this study as determined by the study investigators
* Previous treatment for prostate cancer (surgery, radiotherapy, chemotherapy, hormone androgen deprivation therapy)
* Proven bony metastatic disease, visceral metastases or lymph node metastases above the level of the aortic bifurcation
* Patients who will not get prostatectomy or pelvic lymph node dissection for any reason
* Patient has absolute contra-indications to undergoing MRI scanning

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance between and sensitivity and specificity of PSMA PET-CT and USPIO enhanced MRI | Within 8 weeks before pelvic lymph node dissection
  The sensitivity and specificity of the PSMA PET-CT and nano-MRI will be determined based upon pathological validation

CONTACTS AND LOCATIONS:
Overall Officials: Fred Witjes, PhD, Principal Investigator — Radboud University Medical Centre Nijmegen
Locations (3):
- Netherlands (3):
  - Radboud University Medical Centre, Nijmegen, Gelderland
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Canisius Wilhelmina Ziekenhuis, Nijmegen

IPD SHARING:
Plan to Share IPD: No